CLINICAL TRIAL: NCT06792188
Title: Smartwatch-Based Artificial Intelligence Model for Obstructive Sleep Apnea Prediction
Brief Title: Smartwatch-Based AI Model for OSA Prediction (SWOSA)
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jaeyoung Cho, Associate Professor, Seoul National University Hospital
Other Study IDs: 24111291590
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea of Adult; Screening; Smart Watch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Smart Watch Group: Men and women aged 22 to 85 years who visited Seoul National University Hospital with suspected sleep apnea due to symptoms such as snoring, apnea, or excessive daytime.
  Interventions: Device: Galaxy Watch 4, Samsung Electronics Co., Ltd., South Korea

INTERVENTIONS:
Device: Galaxy Watch 4, Samsung Electronics Co., Ltd., South Korea — Use of the Galaxy Watch 4 during sleep for approximately two weeks prior to the polysomnography test, including the night of the test.

SUMMARY:
This study aims to develop an artificial intelligence (AI) model for more accurately diagnosing obstructive sleep apnea (OSA) by collecting blood oxygen saturation and other health information during sleep using a smartwatch.

OSA is common but often underdiagnosed, and the gold-standard diagnostic test, polysomnography, is costly and time-consuming. Smartwatches can provide a variety of health data, such as sleep patterns, blood oxygen saturation, and heart rate, which can help detect key symptoms and signs of OSA.

By developing an AI model that uses smartwatch data to screen for OSA, this study seeks to offer a cost-effective and accessible diagnostic method, ultimately contributing to the early detection and improved treatment rates of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 22 to 85 years who visited Seoul National University Hospital with suspected sleep apnea due to symptoms such as snoring, apnea, or excessive daytime sleepiness.

Exclusion Criteria:

* Patients previously diagnosed with sleep apnea who are currently undergoing treatment (e.g., positive airway pressure [PAP] therapy, mechanical ventilation, oral appliances, or surgery).
* Patients with neuromuscular diseases or a history of chronic opioid medication use.
* Patients with severe insomnia that is not controlled by medication.
* Patients receiving supplemental oxygen therapy due to underlying conditions such as heart failure, chronic obstructive pulmonary disease, interstitial lung disease, hypoventilation syndrome, or stroke, or whose baseline oxygen saturation is less than 90%.
* Patients with implanted cardiac pacemakers, defibrillators, or other electronic devices.
* Patients inexperienced in using smartphones, apps, or smartwatches.
* Pregnant women.
* Patients unable or unwilling to provide written informed consent.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 22 to 85 years who visited Seoul National University Hospital with suspected sleep apnea due to symptoms such as snoring, apnea, or excessive daytime sleepiness.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive Accuracy of the AI Model for Moderate-to-Severe Obstructive Sleep Apnea | Up to 2 weeks prior to the polysomnography test.
  Evaluation of how well the AI model, developed using clinical data and smartwatch-recorded information including nocturnal oxygen saturation, predicts moderate-to-severe obstructive sleep apnea (defined as apnea-hypopnea index ≥15/hour) diagnosed by polysomnography.

SECONDARY OUTCOMES:
Predictive Accuracy of the Galaxy Watch Sleep Apnea Feature (SAF) | Up to 2 weeks prior to the polysomnography test.
  Assessment of the accuracy of the Galaxy Watch's built-in sleep apnea feature (SAF) in predicting moderate-to-severe obstructive sleep apnea diagnosed by polysomnography.
Comparison of AI Model and Galaxy Watch Sleep Apnea Feature (SAF) Performance | Up to 2 weeks prior to the polysomnography test.
  Comparison of the predictive performance between the AI model developed in this study and the Galaxy Watch's built-in sleep apnea feature (SAF) for detecting moderate-to-severe obstructive sleep apnea.
Comparison of AI Model and STOP-Bang Questionnaire Performance | Up to 2 weeks prior to the polysomnography test.
  Comparison of the predictive performance between the AI model developed in this study and the STOP-Bang questionnaire for detecting moderate-to-severe obstructive sleep apnea.

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyoung Cho, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that support the findings of this study
Supporting Information: Study Protocol